CLINICAL TRIAL: NCT00278200
Title: Vaccination of Patients at High Risk for Post-Transplant Lymphoproliferative Disorder With a Photochemically Inactivated EBV-Infected B-Cell Vaccine
Brief Title: Vaccine Therapy For Patients Being Considered For Organ Transplant Who Are at Risk For PTLD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Loss of funding
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0216; P30CA006973 (NIH); NA_00046066 (Other: JHMIRB)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2019-02

CONDITIONS: Lymphoproliferative Disorder
Keywords: post-transplant lymphoproliferative disorder
MeSH Terms: conditions — Lymphoproliferative Disorders

ARMS (2):
- EBV Seronegative (Experimental): Inactivated EBV-infected vaccine given at Week 0 and Week 4. This arm included all participants who were negative for Epstein-Barr Virus (EBV) at baseline.
  Interventions: Biological: Inactivated EBV-infected vaccine
- EBV Seropositive (Experimental): Inactivated EBV-infected vaccine given at Week 0 and Week 4. This arm included all participants who were positive for Epstein-Barr Virus (EBV) at baseline.
  Interventions: Biological: Inactivated EBV-infected vaccine

INTERVENTIONS:
Biological: Inactivated EBV-infected vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells may help the body build an effective immune response.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy in treating patients who are being considered for solid organ transplant who are at risk for post-transplant lymphoproliferative disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of photochemically-treated autologous Epstein-Barr virus (EBV)-transformed B-lymphoblastoid cell vaccine in generating an EBV-specific T-cell and antibody response in EBV-negative patients or in boosting the response in EBV-positive patients who are being considered for a solid organ transplant and are at high risk for post-transplant lymphoproliferative disorder.
* Determine adverse events associated with this vaccine in these patients.
* Determine the ability of the vaccine to protect from EBV primary infection in EBV-seronegative patients during the time course of the study.

OUTLINE: This is a nonrandomized, pilot study. Patients are stratified according to Epstein-Barr virus (EBV) status (seropositive vs seronegative).

Patients receive photochemically-treated autologous EBV-transformed B-lymphoblastoid cell vaccine intradermally once in weeks 0 and 4.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Being considered for a solid organ transplant
* At high risk for post-transplant lymphoproliferative disorder

PATIENT CHARACTERISTICS:

* Body weight ≥ 25 kg
* Karnofsky performance status 50-100% OR
* Lansky performance status 50-100%
* Not pregnant
* Negative pregnancy test
* Fertile patients must use contraception during and for 2 months after completion of study treatment
* Hemoglobin ≥ 8 g/dL (erythropoietin allowed)
* No history of autoimmune disease, including any of the following:

  * Systemic lupus erythematosus
  * Sarcoidosis
  * Rheumatoid arthritis
  * Glomerulonephritis
  * Vasculitis
* No primary immunodeficiency
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* No corticosteroids for 1 month before and for 1 month after the first study vaccination, except for the following:

  * Physiologic steroid dosing (≤ 20 mg/day of prednisone or steroid equivalent) for adrenal insufficiency
  * Inhaled steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Ambinder, MD, PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject on the EBV seronegative arm was a screen failure. One EBV seronegative subject was not assigned to intervention arm due to physician decision.
  Seven EBV seropositive subjects were not assigned to intervention arm: three due to physician decision; one due to loss of follow-up; one due to death; and two due to subject withdrawal.
Period: Overall Study
Arm/Group | EBV Seronegative | EBV Seropositive
Started | 2 | 12
Completed | 1 | 8
Not Completed | 1 | 4
Not completed — Death | 1 | 3
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- EBV Seronegative: Inactivated EBV-infected vaccine given at Week 0 and Week 4. This arm included all participants who were negative for Epstein-Barr Virus (EBV) at baseline.
  Inactivated EBV-infected vaccine
- EBV Seropositive: Inactivated EBV-infected vaccine given at Week 0 and Week 4. This arm included all participants who were positive for Epstein-Barr Virus (EBV) at baseline.
  Inactivated EBV-infected vaccine
- Total: Total of all reporting groups
Arm/Group | EBV Seronegative | EBV Seropositive | Total
Number analyzed (Participants) | 2 | 12 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 2
  Between 18 and 65 years | 2 | 10 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [18 to 58] | 54 [7 to 64] | 54 [7 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 2 | 4 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 12 | 14

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Vaccine as Assessed by T-cell Responses
Description: Percentage of participants with T-cell responses. For participants who were EBV-seronegative at enrollment, a response is defined as the appearance of EBV-specific T-cells at one month after the second injection. For participants who were EBV-seropositive at enrollment, a response is defined as a two-fold increase over baseline in the frequency of CD8+ T-cells responding to EBV latency antigens at any point during the first 67 days following the first injection.
Time Frame: Up to 67 days
Population: T-cell responses were uninterpretable on lab analysis; therefore, data was not collected to assess this outcome measure.
Arm/Group | EBV Seronegative | EBV Seropositive
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Adverse Events Associated With the Vaccine
Description: Number of participants who received at least one vaccination and experienced at least one grade 3-4 adverse event by CTCAE 2.0 that was attributed to protocol therapy.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | EBV Seronegative | EBV Seropositive
Number analyzed (Participants) | 2 | 12
Participants | 0 | 0

3. Secondary Outcome: Prevention of Primary Epstein-Barr Virus (EBV) Infection
Description: Number of participants who were EBV-seronegative at baseline, received at least one vaccination, subsequently received a solid organ transplant (not part of this protocol), and did not develop a primary EBV infection.
Time Frame: Up to 5 years
Population: Only one participant met the criteria described in the outcome description. This participant was never tested post-transplant for EBV, so no data was collected for this outcome measure.
Arm/Group | EBV Seronegative
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | EBV Seronegative | EBV Seropositive
All-Cause Mortality (participants affected / at risk) | 1/2 | 4/12
Serious Adverse Events (participants affected / at risk) | 1/2 | 2/12
Other Adverse Events (participants affected / at risk) | 1/2 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBV Seronegative (N=2) | EBV Seropositive (N=12)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EBV Seronegative (N=2) | EBV Seropositive (N=12)
Ascites (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bruising (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Cough (General disorders) | 0 (0) | 1 (1)
Diplopia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (2)
Hypertension (General disorders) | 0 (0) | 2 (2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (4) | 5 (15)
Leukopenia (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - unspecified (General disorders) | 0 (0) | 1 (1)
Pain - abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain - axilla (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Gastrointestinal disorders) | 0 (0) | 1 (1)
Streptococcal pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes